CLINICAL TRIAL: NCT07271238
Title: Feasibility Study on the VERAFEYE Imaging and Navigation System for Guided Catheter Ablation Procedures
Acronym: INSiGHT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LUMA Vision Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: INSiGHT-P005
Record Dates: First submitted 2025-11-27; First posted 2025-12-09 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Atrial Fibrillation; Atrial Flutter; Atrial Arrhythmia
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atrial Fibrillation and Atrial Flutter arm (Experimental): Subjects entitled to undergo a catheter-based ablation treatment for typical atrial flutter and/or atrial fibrillation
  Interventions: Device: VERAFEYE Imaging and Guidance System

INTERVENTIONS:
Device: VERAFEYE Imaging and Guidance System — The VERAFEYE Imaging and Guidance System will be used during standard of care, catheter-based treatments for atrial flutter and/or atrial fibrillation.

SUMMARY:
The objective of the study is to collect data on the usability and integration of the VERAFEYE Imaging and Guidance System in adult patients indicated to undergo a standard of care catheter-based ablation procedure for the treatment of Atrial Flutter (AFL), paroxysmal AF (PAF) or persistent AF (perAF).

Results from this study may be used to guide development and refinement the VERAFEYE Imaging and Guidance System capabilities.

ELIGIBILITY:
Inclusion Criteria:

* IC1: Subject is at least 18 years of age at the time of consent
* IC2: Subject is scheduled to undergo a standard of care catheter-ablation procedure to treat AFL/AF, according to current international and local guidelines and per physician discretion
* IC3: Subject is able to understand and willing to provide written informed consent
* IC4: Subject is able and willing to complete all study assessments associated with this clinical study at an approved clinical study site

Exclusion Criteria:

* EC1: Subject where placement of VERAFEYE Imaging Catheter is technically not feasible per physician discretion
* EC2: Pregnant women or women who plan to become pregnant during the course of their participation in the study (women should either be of non- childbearing potential at the time of enrolment (as documented in the medical file) or have a negative pregnancy test within the previous 7 days prior to the procedure)
* EC3: Subject implanted with an active cardiac rhythm management device (e.g. pacemaker, CRT, ICD)
* EC4: Unrecovered/unresolved Adverse Events from any previous invasive procedure
* EC5: Any planned surgical or endovascular intervention within 30 days before or after the ablation procedure
* EC6: Life expectancy less than 12 months
* EC7: Current LA thrombus Note: Screening for LA thrombus is required to be performed within 48 hours prior to or during the index procedure. Method of screening per physician discretion. If an atrial thrombus is observed prior to or during the planned index procedure, the index procedure will not begin or will be terminated before accessing the left atrium, and no ablation will be performed. The index procedure for this subject may be rescheduled to be performed within 30 days post ICF signature, provided that the thrombus is no longer present.
* EC8: Subjects who are currently enrolled in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
ADEs | within 7 days of the index procedure
  • Rate of device-related adverse events (ADEs) occurring within 7 days of the index procedure
VERAFEYE Performance | during procedure
  • Ability of VERAFEYE Imaging and Guidance System to:
  * Visualize major cardiac structures (e.g. RA, septum, LA, PVs)
  * Create 3D anatomical model with the VERAFEYE Imaging and Guidance System